CLINICAL TRIAL: NCT04635293
Title: Preoperative Infusion of Levosimendan in High Risk Cardiac Surgery Patients: A Retrospective Study
Brief Title: Preoperative Infusion of Levosimendan in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 667/24.02.2020
Record Dates: First submitted 2020-11-09; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Disease; Cardiac Failure; Cardiac Surgery; Inotropes; Ejection Fraction
Keywords: levosimendan; low output syndrome
MeSH Terms: conditions — Heart Diseases; Heart Failure

STUDY DESIGN:
Intervention Model Description: Retrospective
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients who were administered levosimendan at a dose of 0.1µg/Kg/min for 24 hours prior to surgery (Active Comparator)
  Interventions: Procedure: preoperative infusion of levosimendan
- patients who were not administered levosimendan prior to surgery (Placebo Comparator)
  Interventions: Procedure: no preoperative infusion of levosimendan

INTERVENTIONS:
Procedure: preoperative infusion of levosimendan — the study group will consist of patients who have received a continuous infusion of levosimendan 0.1 μg/kg/min for 24 hours before cardiac surgery
  Arms: patients who were administered levosimendan at a dose of 0.1µg/Kg/min for 24 hours prior to surgery
Procedure: no preoperative infusion of levosimendan — the control group will consist of patients who proceeded to the cardiac operation without any infusion for 24 hours preoperatively
  Arms: patients who were not administered levosimendan prior to surgery

SUMMARY:
The aim of this retrospective study will be to investigate the effect of the preoperative administration of levosimendan on the outcome of patients with compromised cardiac function undergoing cardiac surgery

DETAILED DESCRIPTION:
Patients with severely reduced left ventricular ejection fraction (LVEF) face a high risk of morbidity and mortality after cardiac surgery. Impaired cardiac function preoperatively predisposes patients to low cardiac output syndrome. Levosimendan acts by a different mechanism than traditional inotropes and its preoperative use could improve the outcome of patients with cardiac failure. Specifically, it promotes vasodilation of coronary, pulmonary and systemic vessels, has an anti-inflammatory and anti-oxidant effect and enhances cardiac contractility by improving the response of the myofilaments to intracellular calcium.

The aim of this retrospective study will be to investigate the effect of the preoperative administration of levosimendan on the outcome of patients with compromised cardiac function undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery
* cardiac surgery under cardiopulmonary bypass
* low ejection fraction (<40%)

Exclusion Criteria:

* age <18 years old
* urgent operation
* glomerular filtration rate<30 ml/min
* hepatic dysfunction preoperatively
* side effects (hypotension, tachycardia, ST segment abnormalities during levosimendan administration
* redo surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
hours of mechanical ventilation | during stay in ICU, approximately 48 hours postoperatively
  hours of mechanical ventilation during patient stay in Intensive Care Unit (ICU)
vasopressor use in operating room | intraoperatively, from induction to end of anesthesia, an average period of 3 hours
  need for vasopressor use, yes or no
vasopressor use in ICU | during stay in ICU, approximately 48 hours postoperatively
  need for vasopressor use, yes or no
inotrope use in operating room | intraoperatively, from induction to end of anesthesia, an average period of 3 hours
  need for inotrope use, yes or no
inotrope use in ICU | during stay in ICU, approximately 48 hours postoperatively
  need for inotrope use, yes or no
incidence of arrhythmias | postoperatively, an average period of 7-10 days
  development of new-onset arrhythmias, yes or no
incidence of renal dysfunction | postoperatively, an average period of 7-10 days
  development of new-onset renal dysfunction, defined as an increase in creatinine levels over 0.3 mg/dL from the initial values
length of ICU stay | postoperatively, an average period of 7-10 days
  duration of patient stay in ICU in days
hospitalization time | postoperatively, up to 20 days after the operation
  duration of hospital stay after surgery in days
incidence of death within the first 30 days after surgery | 30 days after surgery
  patient survival within the first 30 days after surgery, yes or no
need of mechanical assist devices intraoperatively | intraoperatively, from induction to end of anesthesia, an average period of 3 hours and postoperatively, an average period of 7-10 days
  need for mechanical assist devices, yes or no
need of mechanical assist devices postoperatively | postoperatively, an average period of 7-10 days
  need for mechanical assist devices, yes or no
change from baseline in cardiac output (CO) | 10 minutes after anesthesia induction, 10 minutes after bypass discontinuation, end of operation (an average period of 3 hours after start of surgery), 12 hours after ICU admittance, 24 hours after ICU admittance,
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in mean arterial pressure (MAP) | 10 minutes after anesthesia induction, 10 minutes after bypass discontinuation, end of operation (an average period of 3 hours after start of surgery), 12 hours after ICU admittance, 24 hours after ICU admittance,
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in mean pulmonary arterial pressure (MPAP) | 10 minutes after anesthesia induction, 10 minutes after bypass discontinuation, end of operation (an average period of 3 hours after start of surgery), 12 hours after ICU admittance, 24 hours after ICU admittance,
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in systemic vascular resistance (SVR) | 10 minutes after anesthesia induction, 10 minutes after bypass discontinuation, end of operation (an average period of 3 hours after start of surgery), 12 hours after ICU admittance, 24 hours after ICU admittance,
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in pulmonary vascular resistance (PVR) | 10 minutes after anesthesia induction, 10 minutes after bypass discontinuation, end of operation (an average period of 3 hours after start of surgery), 12 hours after ICU admittance, 24 hours after ICU admittance,
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in pulmonary capillary wedge pressure (PCWP) | 10 minutes after anesthesia induction, 10 minutes after bypass discontinuation, end of operation (an average period of 3 hours after start of surgery),12 hours after ICU admittance, 24 hours after ICU admittance,
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in cardiac function | 10 minutes after anesthesia induction, 10 minutes after bypass discontinuation, end of operation (an average period of 3 hours after start of surgery)
  transesophageal echocardiography will be used for echocardiographic measurements

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Onassis Cardiac Surgery Center, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tasouli A, Papadopoulos K, Antoniou T, Kriaras I, Stavridis G, Degiannis D, Geroulanos S. Efficacy and safety of perioperative infusion of levosimendan in patients with compromised cardiac function undergoing open-heart surgery: importance of early use. Eur J Cardiothorac Surg. 2007 Oct;32(4):629-33. doi: 10.1016/j.ejcts.2007.07.010. Epub 2007 Aug 15. PMID 17702589
- [Background] Landoni G, Biondi-Zoccai G, Greco M, Greco T, Bignami E, Morelli A, Guarracino F, Zangrillo A. Effects of levosimendan on mortality and hospitalization. A meta-analysis of randomized controlled studies. Crit Care Med. 2012 Feb;40(2):634-46. doi: 10.1097/CCM.0b013e318232962a. PMID 21963578
- [Background] Tritapepe L, De Santis V, Vitale D, Guarracino F, Pellegrini F, Pietropaoli P, Singer M. Levosimendan pre-treatment improves outcomes in patients undergoing coronary artery bypass graft surgery. Br J Anaesth. 2009 Feb;102(2):198-204. doi: 10.1093/bja/aen367. PMID 19151048
- [Background] De Hert SG, Lorsomradee S, Cromheecke S, Van der Linden PJ. The effects of levosimendan in cardiac surgery patients with poor left ventricular function. Anesth Analg. 2007 Apr;104(4):766-73. doi: 10.1213/01.ane.0000256863.92050.d3. PMID 17377079
- [Background] Kivikko M, Lehtonen L. Levosimendan: a new inodilatory drug for the treatment of decompensated heart failure. Curr Pharm Des. 2005;11(4):435-55. doi: 10.2174/1381612053382043. PMID 15725064
- [Background] Mehta RH, Leimberger JD, van Diepen S, Meza J, Wang A, Jankowich R, Harrison RW, Hay D, Fremes S, Duncan A, Soltesz EG, Luber J, Park S, Argenziano M, Murphy E, Marcel R, Kalavrouziotis D, Nagpal D, Bozinovski J, Toller W, Heringlake M, Goodman SG, Levy JH, Harrington RA, Anstrom KJ, Alexander JH; LEVO-CTS Investigators. Levosimendan in Patients with Left Ventricular Dysfunction Undergoing Cardiac Surgery. N Engl J Med. 2017 May 25;376(21):2032-2042. doi: 10.1056/NEJMoa1616218. Epub 2017 Mar 19. PMID 28316276
- [Background] Cholley B, Caruba T, Grosjean S, Amour J, Ouattara A, Villacorta J, Miguet B, Guinet P, Levy F, Squara P, Ait Hamou N, Carillion A, Boyer J, Boughenou MF, Rosier S, Robin E, Radutoiu M, Durand M, Guidon C, Desebbe O, Charles-Nelson A, Menasche P, Rozec B, Girard C, Fellahi JL, Pirracchio R, Chatellier G; -. Effect of Levosimendan on Low Cardiac Output Syndrome in Patients With Low Ejection Fraction Undergoing Coronary Artery Bypass Grafting With Cardiopulmonary Bypass: The LICORN Randomized Clinical Trial. JAMA. 2017 Aug 8;318(6):548-556. doi: 10.1001/jama.2017.9973. PMID 28787507
- [Background] Papp Z, Edes I, Fruhwald S, De Hert SG, Salmenpera M, Leppikangas H, Mebazaa A, Landoni G, Grossini E, Caimmi P, Morelli A, Guarracino F, Schwinger RH, Meyer S, Algotsson L, Wikstrom BG, Jorgensen K, Filippatos G, Parissis JT, Gonzalez MJ, Parkhomenko A, Yilmaz MB, Kivikko M, Pollesello P, Follath F. Levosimendan: molecular mechanisms and clinical implications: consensus of experts on the mechanisms of action of levosimendan. Int J Cardiol. 2012 Aug 23;159(2):82-7. doi: 10.1016/j.ijcard.2011.07.022. Epub 2011 Jul 23. PMID 21784540